CLINICAL TRIAL: NCT00289848
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Study of MK0431 in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control
Brief Title: MK0431 Monotherapy Study in Patients With Type 2 Diabetes Mellitus (0431-040)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-040; MK0431-040; 2005_094
Record Dates: First submitted 2006-02-07; First posted 2006-02-10 (Estimated); Results first posted 2010-04-02 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): sitagliptin 100 mg
  Interventions: Drug: sitagliptin phosphate
- 2 (Placebo Comparator): placebo
  Interventions: Drug: Comparator: placebo

INTERVENTIONS:
Drug: sitagliptin phosphate — Sitagliptin 100 mg administered as one oral tablet once daily before the morning meal for up to 18 weeks.
  Other Names: Januvia
  Arms: 1
Drug: Comparator: placebo — placebo to match Sitagliptin 100 mg administered as one oral tablet once daily before the morning meal for up to 18 weeks
  Arms: 2

SUMMARY:
This is a clinical study to determine the safety and efficacy of an investigational drug in patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Patients have Type 2 Diabetes Mellitus and have laboratory results that are within the values established by the study such as an Hemoglobin A1c (HbA1c) >=7.5% and <=11% and a Fasting Plasma Glucose (FPG) >=130 mg/dL and <=280 mg/dL

Exclusion Criteria :

* Patients have Type 1 Diabetes Mellitus or required insulin therapy within the past 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2006-03; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Mohan V, Yang W, Son HY, Xu L, Noble L, Langdon RB, Amatruda JM, Stein PP, Kaufman KD. Efficacy and safety of sitagliptin in the treatment of patients with type 2 diabetes in China, India, and Korea. Diabetes Res Clin Pract. 2009 Jan;83(1):106-16. doi: 10.1016/j.diabres.2008.10.009. Epub 2008 Dec 20. PMID 19097665
- [Derived] Singh B, Sims H, Trueheart I, Simpson K, Wang KC, Patzkowsky K, Wegman T, Soma JM, Dixon R, Jayes F, Voegltine K, Yenokyan G, Su SC, Leppert P, Segars JH. A Phase I Clinical Trial to Assess Safety and Tolerability of Injectable Collagenase in Women with Symptomatic Uterine Fibroids. Reprod Sci. 2021 Sep;28(9):2699-2709. doi: 10.1007/s43032-021-00573-8. Epub 2021 Apr 29. PMID 33914296

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In: 27-Apr-2006; Last Patient Last Visit: 30-Mar-2007; Twenty-eight medical clinics (9 in China, 9 in India, and 10 in Korea).
Pre-assignment Details: Patients not on an antihyperglycemic agent (AHA) or on oral single AHA or low dose dual combination therapy could participate. After an up to 6-week diet/exercise (and wash-off period for patients on AHA), patients with hemoglobin A1C 7.5-11% and fasting plasma glucose 130-280 mg/dL entered a 2-week placebo run-in period prior to randomization.
Groups:
- Sitagliptin 100 mg: The Sitagliptin 100 mg group includes data from patients randomized to receive treatment with 100 mg oral tablets of sitagliptin once daily.
- Placebo: The Placebo group includes data from patients randomized to receive treatment with oral tablets of sitagliptin-matching placebo once daily.
Period: Overall Study
Arm/Group | Sitagliptin 100 mg | Placebo
Started | 352 | 178
Completed | 306 | 133
Not Completed | 46 | 45
Not completed — Adverse Event | 6 | 4
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 20 | 24
Not completed — Lost to Follow-up | 3 | 1
Not completed — Protocol Violation | 5 | 2
Not completed — Withdrawal by Subject | 5 | 11
Not completed — Patient Moved | 6 | 2
Not completed — Open-Label AHA Treatment Requested | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin 100 mg | Placebo | Total
Number analyzed (Participants) | 352 | 178 | 530
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (9.3) | 50.9 (9.3) | 50.9 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 72 | 224
  Male | 200 | 106 | 306
Race/Ethnicity, Customized [Number; unit: participants]
  Chinese | 163 | 82 | 245
  Indian | 127 | 63 | 190
  Korean | 62 | 33 | 95
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 189.0 (44.0) | 190.2 (46.2) | 189.4 (44.7)
Hemoglobin A1C (HbA1C; A1C) [Mean (Standard Deviation); unit: Percent] | 8.74 (1.01) | 8.75 (1.06) | 8.74 (1.03)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at Week 18
Description: A1C was measured as a percent. Thus, this change from baseline reflects the Week 18 A1C percent minus the Week 0 A1C percent.
Time Frame: Baseline and Week 18
Population: The full-analysis-set (FAS) population included all patients with at least one dose of double-blind study therapy, and with a baseline value and ≥1 post-baseline value for this outcome. Missing data were handled using the last observation carrying forward (LOCF) method.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 339 | 169
Percent | -0.71 [-0.84 to -0.59] | 0.31 [0.14 to 0.48]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA with terms of treatment, country, prior diabetes pharmacotherapy (not on AHA or on AHA), and baseline A1C as a covariate; Mean Difference (Net) = -1.03, 95% CI [-1.23 to -0.83], Standard Deviation 1.08

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 18
Description: Change from baseline at Week 18 is defined as Week 18 FPG minus Week 0 FPG.
Time Frame: Baseline and Week 18
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 339 | 169
mg/dL | -25.8 [-30.3 to -21.3] | 5.2 [-1.0 to 11.4]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA with terms of treatment, country, prior diabetes pharmacotherapy (not on AHA or on AHA), and baseline FPG as a covariate; Mean Difference (Net) = -31.0, 95% CI [-38.4 to -23.7], Standard Deviation 39.8

3. Secondary Outcome: Change From Baseline in 2-hr Post-Meal Glucose (PMG) at Week 18
Description: Change from baseline at Week 18 is defined as Week 18 minus Week 0.
Time Frame: Baseline and Week 18
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 297 | 131
mg/dL | -63.8 [-71.0 to -56.6] | -7.2 [-17.7 to 3.3]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA with terms of treatment, country, prior diabetes pharmacotherapy (not on AHA or on AHA), and baseline 2-hr PMG as a covariate; Mean Difference (Net) = -56.6, 95% CI [-68.8 to -44.3], Standard Deviation 59.2

ADVERSE EVENTS:
Arm/Group | Sitagliptin 100 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 6/352 | 2/178
Other Adverse Events (participants affected / at risk) | 0/352 | 0/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin 100 mg (N=352) | Placebo (N=178)
Any Cardiac Disorders (Cardiac disorders) | 1 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 0
Myocardial Ischaemia (Cardiac disorders) | 0 | 1
Any Hepatobiliary Disorders (Hepatobiliary disorders) | 1 | 0
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0
Any Neoplasms Benign, Malignant And Unspecified (Incl Cysts & Polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Carcinoid Tumour Of The Gastrointestinal Tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian Epithelial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Any Nervous System Disorders (Nervous system disorders) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Any Psychiatric Disorders (Psychiatric disorders) | 0 | 1
Alcoholism (Psychiatric disorders) | 0 | 1
Any Respiratory, Thoracic And Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.